CLINICAL TRIAL: NCT02562534
Title: Use of a New ElectroCardioGraph to Create an ECG Database in 3T MRI With Healthy Heart and Several Kind of Cardiac Disease in Order to Let go of Artifacts.
Brief Title: Creation of an ECG Database in 3T MRI With Healthy Heart and Several Kind of Cardiac Disease.
Acronym: DB-ECG-3T
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was sufficient data to verify the primary endpoint
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Jean-Marc SELLAL, Cardiologist specialised in rhythmology, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A01406-37
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Heart Diseases
Keywords: ECG; MRI; rhythm troubles; conductive troubles; ECG artifacts; Database
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with conductive troubles (Other): Patients with conductive troubles
  Interventions: Device: MRI compatible ElectroCardioGraph
- Patients with rhythm troubles (Other): Patients with rhythm troubles
  Interventions: Device: MRI compatible ElectroCardioGraph
- Volunteers (Other): Volunteers with normal ECG
  Interventions: Device: MRI compatible ElectroCardioGraph

INTERVENTIONS:
Device: MRI compatible ElectroCardioGraph — MRI with ECG control for people with healthy heart or heart diseases

SUMMARY:
The aim is to create a database including recordings of ECG data recorded in an MRI acquisition

DETAILED DESCRIPTION:
ECG monitoring is an essential tool during MRI, especially for cardiac MRI (CMR). Indeed, the system needs to synchronize the acquisitions on the cardiac cycles. To identify the cycle, the system is based on the ECG. Furthermore, patients having a CMR can be at risk of presenting cardiac rhythm troubles, and must be monitored with a trustable system.

The problem is that in MRI, a lot of artefacts occur, leading to dramatic disturbances of the signal. A lot of tools are used to try to remove the artefacts. The aim of this study is to create a database that can be used to test the different tools to remove the artefacts.

The investigators intend to include all types of ECG patterns that can exist, to allow to test the tools in all situations.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects:

  * To be more than 18
  * To be enroled in a social security plan
  * To have signed an informed consent
  * To have preliminary medical examination
* For the groups :

  * "normal ECG" group : sinus rhythm without conductive troubles. Normal pattern of the QRS
  * "conductive troubles group" : patients with typical right bundle branch block, or typical left bundle branch block pattern.
  * "rhythm trouble group" : patients with premature atrial beats or premature ventricular beats

Exclusion Criteria:

* Contraindication: implantable devices (cardiac stimulators, defibrillators, cochlear implants, etc.), metallic foreign bodies
* Impossibility to undergo MRI: claustrophobia, morbid obesity.
* Pregnancy or risk of pregnancy.
* Patients under a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the ECG signal quality | One year
  Evaluation of the ECG signal quality acquired in the MRI 3 Tesla by measuring the amplitude of the QRS complex (in millivolts). Conformity with IEC (International Electrotechnical Commission) 60601-2-51 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Chillou, Pr, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Universitaire de Nancy, Nancy, France